CLINICAL TRIAL: NCT05719064
Title: Adaptive Cell Phone Support to Promote Medication Adherence Among Adolescents and Young Adults With Chronic Health Conditions
Brief Title: Early Prototyping and Usability Testing (ACPS)
Acronym: ACPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Caitlin Sayegh, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-23-00149_Phase I
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Medication Adherence
Keywords: Adolescents; Mobile health; chronic illness
MeSH Terms: conditions — Medication Adherence; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adaptive Cell Phone Support (Experimental): Computer-delivered cell phone support (reminders, problem-solving, referrals to resources) and responsive human coaching (phone calls, test messages, in-app messaging) to improved medication adherence.
  Interventions: Behavioral: Adaptive Cell Phone Support

INTERVENTIONS:
Behavioral: Adaptive Cell Phone Support — Mobile health adherence promotion based on the supportive accountability model

SUMMARY:
The goal of this pilot clinical trial is to refine and test a mobile health intervention for promoting medication adherence in a population of adolescents and young adults with chronic health conditions. The main question[s] it aims to answer are:

* How should the intervention be designed to best fit patients' needs and preferences?
* Is an adaptive intervention (personalizing the intensity of support based on patients' needs) efficacious for promoting medication adherence Researchers will compare the adaptive intervention to automated text message reminders see if the adaptive intervention shows stronger positive effects on medication adherence.

DETAILED DESCRIPTION:
An initial cohort of adolescents with chronic health conditions will be asked to try the intervention and give feedback to refine the structure and content. Then, a larger cohort will progress through a sequential multiple assignment randomized trial to 1) be randomized to either automated text reminders (active control condition) or computer-delivered Cell Phone Support and then 2) those in the computer-delivered Cell Phone Support condition who do not show a sufficient response will be re-assigned to continued computer-delivered Cell Phone Support only or to Adaptive Cell Phone Support ( computer-delivered Cell Phone Support + responsive human coaching).

ELIGIBILITY:
Inclusion Criteria:

* Children's Hospital Los Angeles patient
* between 15-20 years old
* taking at least one oral medication per day for a chronic health condition
* English speaking
* demonstrating sufficient cognitive capacity to engage in the assent/consent process and study procedures
* has a cell phone

There is no exclusion criteria.

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Mean scores on the Mobile Health App Usability Questionnaire | Baseline to 3 weeks
  Higher scores indicate greater ease with which users can use technology to achieve a particular goal; the minimum value of this questionnaire is 1 and the maximum value is 7.
Total scores on the theoretical framework of acceptability questionnaire | Baseline to 3 weeks
  Higher scores indicate a greater "extent to which people delivering or receiving a healthcare intervention consider it to be appropriate, based on anticipated or experienced cognitive and emotional responses to the intervention"; the minimum value of this questionnaire is 7 and the maximum value is 35.
Total scores on the Visual Analogue Scale | Baseline to 3 weeks
  Percentage of doses taken our of 100%; higher numbers indicate greater medication adherence. This scale presents participants with a line, marked 0 on the left and 100 on the right, and participants can drag a marker to the place on the line that best visually indicated their adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Sayegh, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data and associated documentation will be made available to the research community free of charge through the data repository hosted at Open Science Framework (OSF).
Time Frame: Final submission and release of the study data will occur within 12 months of the conclusion of data collection, and within the award period. Study data deposited in OSF will be available to the research community in perpetuity.
Access Criteria: Any OSF users can access the de-identified data.
URL: https://osf.io/